CLINICAL TRIAL: NCT06216106
Title: Prepectoral Breast Reconstruction With Polyurethane Implantes and Radiotherapy: a Single Center Retrospective Study Evaluating Risk and Complications
Brief Title: Data Collection of Prepectoral Breast Reconstruction With Polyurethane Implantes
Acronym: IBR-PPBR
Status: Completed | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 4260
Record Dates: First submitted 2023-12-21; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-09

CONDITIONS: Prepectoral Breast Reconstruction; Breast Reconstruction; Radiation Therapy Complication
Keywords: PPBR; POLYURETHANE; IBR; RADIOTHERAPY; BREAST IMPLANTS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients undergone prepectoral breast reconstruction: As the retrospective nature of this study, we have no exlusion criterias. We included all the patients with prepectoral breast reconstruction with polyurethane covered implants. We also included patients underwent postoperative radiation therapy (50 patients) and 20 patients with history of previous radiotherapy
  Interventions: Procedure: Prepectoral breast reconstruction with polyurethane implants

INTERVENTIONS:
Procedure: Prepectoral breast reconstruction with polyurethane implants — Breast reconstruction in the prepectoral plane without elevate the pectoralis major muscle. We choose this type of reconstruction only in patients with mastectomy flap thickness of plus then 0.5 cm. We usally use silicone implants covered by an external layer of polyurethane so not to put directly in contact the silicone with the subcutaneus tissue.

SUMMARY:
The goal of this observational study is to learn about correct surgical indications and long-term complications in patient with immediate prepectoral breast reconstruction with polyurethane implants. The main question it aims to answer are: what are the correct indications for this type of reconstruction? what is the complications rates? are the complications affected by pre and post operative radiotherapy? It's a retrospective study of all the patients that received prepectoral breast reconstruction with polyurethane implants without any exclusion factors. Researchers will compare the non-irradiated group with the patients with pre and post radiation therapy.

DETAILED DESCRIPTION:
The study is a data collection of 250 patients for a total of 317 breasts underwent prepectoral breast recosntruction with polyurethane implantes. It is a retrospective study of a single center. The investigators gave indication to that type of reconstruction only to patients with good thickness (> 0.5 cm) and vascularity of skin flap after mastectomy.

The investigators used not selective criteria regarding risk factors so to better evaluate wich of them has a negative trend on the success of the reconstruction and on the major and minor complications. In that way the investigators tried to definde clarly the correct indications for this type of reconstruction.

In addition, the investigators would like to define if the postoperative radiation therapy agument the complications rate and the capsular contracture incidence.

The investigators decide to perform prepectoral breast reconstruction also in 20 patientes underwent previous radiotherapy dependig on the grade of cutaneus radiodistrophy, so to propose our less invasive approach to these patients normally candidates to autologus breast reconstruction

ELIGIBILITY:
Inclusion Criteria:

* patients underwent prepectoral breast recosntruction with polyurethane implants after skin or nipple sparing masectomy
* adequate mastectomy flap in vascularity and thickness

Exclusion Criteria:

* none

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — we included only famale patients underwent mastectomy and immediate breast reconstruction in the prepectoral plane with polyurethane implantes
Study Population: Patientes undergone immediate prepectoral breast reconstruction with polyurethane implantes
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
reconstruction failure | 12 months
  loss of implant or switch to autologus recosntruction
major complications | 12months
  evaluation of hematoma, infection, flap necrosis, wound dehiscence rate
minor complications | 12 months
  evaluation of seroma, rippling, casular contracture, asymmetry rate
risk factor | 12 months
  evaluation of the risk factors correlated to recostruction failure

SECONDARY OUTCOMES:
postoperative radiation therapy on patients underwent prepectoral breast reconstruction with polyurethane implantes | 12 months
  evaluation if the post operative radiation therapy is correlated with an increase of reconstruction failure and capsular contracture
patients previously irradiated (QUART) and underwent prepectoral breast reconstruction with polyurethane implantes | 12 months
  analysis of clinical characteristics of pre irradiatred patients submitted to prepectoral breast recosntruction with polyurethane implantes

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Vittorio Emanuele Lisa, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- European Institute of Oncology, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salgarello M, Pagliara D, Barone Adesi L, Visconti G, Wild JB, Matey P. Direct to Implant Breast Reconstruction With Prepectoral Micropolyurethane Foam-Coated Implant: Analysis of Patient Satisfaction. Clin Breast Cancer. 2021 Aug;21(4):e454-e461. doi: 10.1016/j.clbc.2021.01.015. Epub 2021 Jan 23. PMID 33627298
- [Background] de Vita R, Buccheri EM, Villanucci A, Pozzi M. Breast Reconstruction Actualized in Nipple-sparing Mastectomy and Direct-to-implant, Prepectoral Polyurethane Positioning: Early Experience and Preliminary Results. Clin Breast Cancer. 2019 Apr;19(2):e358-e363. doi: 10.1016/j.clbc.2018.12.015. Epub 2018 Dec 27. PMID 30691930